CLINICAL TRIAL: NCT02333175
Title: Care for Late Stage Parkinsonism
Acronym: CLaSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Philipps University Marburg (Other); Instituto de Medicina Molecular João Lobo Antunes (Other); University Medical Center Nijmegen (Other); Lund University (Other); University Hospital, Bordeaux (Other); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14/0040
Record Dates: First submitted 2014-09-25; First posted 2015-01-07 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Parkinson's Disease; Late Stage Parkinson's Disease
Keywords: Parkinson's disease, Late stage
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Specialist review (Active Comparator): Specialist review with individually tailored treatment strategies suggested by specialist
  Interventions: Other: Specialist review
- Care as usual (No Intervention): Care as usual

INTERVENTIONS:
Other: Specialist review — Specialist review with individually tailored treatment strategies suggested by specialist
  Arms: Specialist review

SUMMARY:
The aim of this project is to evaluate the needs and provision of care for patients in the late stages of Parkinsonism and their carers in several European countries, to compare the effectiveness of different health and social care systems, and to lay the foundation for improved outcomes in this population. The investigators will undertake an in-depth assessment of patients and their care arrangements in a population recruited through networks in six European countries. The systems and procedures that are used in the provision of care will be reviewed through a systematic literature review, interviews and assessments of patients, carers and health care providers, and through a trial comparing assessment by a specialist with management suggestions, guidance and access to telephone advice to that of usual care. Through interviews, questionnaire assessment and review of current health-care and social care arrangement, the investigators will assess the needs, provision of care and use of health-care resources, and their impact on patient and carer outcomes in different countries. National and regional databases will also be interrogated to identify current practice and use of healthcare resources and drug usage. A systematic literature review of the evidence for effective management strategies, analysis of the study data, and evaluation of change in outcomes following specialist review will provide the basis for recommendations in the management of late stage Parkinsonism. The investigators will also evaluate potentially useful outcome measures for use in this patient group. In addition to charting the needs and current care provision for late stage Parkinsonism in different European countries, its cost and effectiveness, and an analysis of health-care and social care predictors of improved outcome, the project will produce a platform for the assessment of patients with late stage Parkinsonism, their current treatment and care provision, as well as guidelines on the management of this late disease phase.

ELIGIBILITY:
Inclusion Criteria:

* Hoehn and Yahr stage (HY) IV or V in the "On"-state
* Disease duration of at least 7 years

Exclusion Criteria:

* Symptomatic Parkinsonism

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
UPDRS-ADL part | 6 months
  Disability measure

SECONDARY OUTCOMES:
PDQ-8 or DEMQoL proxy | 6 months
  Quality of Life
Zarit carer burden scale | 6 months
  Carer burden
Satisfaction with care Likert scale | 6 months
MMSE | 6 months
  Mental health
NPI | 6 months
  Mental health
UPDRS III | 6 months
  PD severity
NMSS | 6 months
  PD severity
PD milestones | 6 months
  PD severity
Basic palliative care assessment | 6 months
  ESAS-PD

CONTACTS AND LOCATIONS:
Locations (7):
- University of Bordeaux, Bordeaux, France
- Germany (2):
  - University of Munich, Munich, Bavaria
  - University of Marburg, Marburg
- Radboud university medical center, Nijmegen, Netherlands
- Instituto de Medicina Molecular, Lisbon, Portugal
- Lund University, Lund, Sweden
- University College London, London, United Kingdom

REFERENCES:
- [Derived] Kruse C, Kretschmer S, Lipinski A, Verheyen M, Mengel D, Balzer-Geldsetzer M, Lorenzl S, Richinger C, Schmotz C, Tonges L, Woitalla D, Klebe S, Schrag A, Dodel R. Resource Utilization of Patients with Parkinson's Disease in the Late Stages of the Disease in Germany: Data from the CLaSP Study. Pharmacoeconomics. 2021 May;39(5):601-615. doi: 10.1007/s40273-021-01011-y. Epub 2021 Mar 19. PMID 33738776
- [Derived] Balzer-Geldsetzer M, Ferreira J, Odin P, Bloem BR, Meissner WG, Lorenzl S, Wittenberg M, Dodel R, Schrag A. Study protocol: Care of Late-Stage Parkinsonism (CLaSP): a longitudinal cohort study. BMC Neurol. 2018 Nov 5;18(1):185. doi: 10.1186/s12883-018-1184-3. PMID 30396331